CLINICAL TRIAL: NCT01591655
Title: The Efficacy and Safety of Mapracorat Ophthalmic Suspension, 3% in Subjects for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery.
Brief Title: Mapracorat Ophthalmic Suspension, 3% for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 793
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Cataract; Inflammation; Surgery
MeSH Terms: conditions — Cataract; Inflammation | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mapracorat (Experimental): Mapracorat ophthalmic suspension, 3%,
  Interventions: Drug: Mapracorat
- Vehicle (Placebo Comparator): The vehicle of the mapracorat ophthalmic suspension
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Mapracorat — 1 drop of study medication into the study eye four times daily (QID) for 14 days
  Arms: Mapracorat
Drug: Vehicle — 1 drop of vehicle into the study eye QID for 14 days.
  Arms: Vehicle

SUMMARY:
The objective of this clinical study is to compare the safety and efficacy of mapracorat ophthalmic suspension, 3% with its vehicle for the treatment of postoperative inflammation and pain following cataract surgery. Participants from the United States and Canada will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are candidates for routine, uncomplicated cataract surgery.
* Subjects who, in the Investigator's opinion, have potential postoperative pinhole Snellen visual acuity (VA) of at least 20/200 in the study eye.
* Subjects who have ≥ Grade 2 (6 - 15 cells) AC cells in the study eye following cataract surgery (postoperative day 1).

Exclusion Criteria:

* Subjects who have a severe/serious ocular condition or history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result(s) of the study.
* Any intraocular inflammation in either eye (cells or flare score greater than Grade 0 at slit lamp examination) or ocular pain greater than Grade 1 in the study eye at the Screening Visit.
* Presence of active external ocular disease: infection or inflammation of the study eye.
* Subjects who have known hypersensitivity or contraindication to the study drug(s) or their components.
* Subjects who currently require or are expected to require treatment with any medication listed as a disallowed medication per the Disallowed Therapy section of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quintus Ngumah, OD,PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mapracorat | Vehicle
Started | 240 | 120
Completed | 168 | 57
Not Completed | 72 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mapracorat | Vehicle | Total
Number analyzed (Participants) | 240 | 120 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (10.27) | 67.4 (8.59) | 67.2 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 67 | 204
  Male | 103 | 53 | 156

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells
Description: Anterior chamber (AC) cells were assessed using a 0 to 4 grading scale by an ophthalmologist using slip lamp biomicroscopy. A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens was performed without pupil dilation. Accumulation of white blood cells in aqueous was assessed. The grades were defined as: 0 = No cells seen; 1 = 1 - 5 cells; 2 = 6 - 15 cells; 3 = 16 - 30 cells; 4 = >30 cells. Complete resolution of AC cells was defined as Grade 0.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 240 | 120
Participants | 38 | 13

2. Primary Outcome: Percentage of Participants With Grade 0 Pain
Description: Ocular pain was defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching. The scores ranged from 0=None to 5=Severe, where higher scores indicated worse pain.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 240 | 120
Participants | 172 | 59

3. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells.
Description: as for outcome 1
Time Frame: 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 240 | 120
Participants | 71 | 21

4. Secondary Outcome: Percentage of Participants With Grade 0 Pain
Description: Ocular pain was defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching. The scores ranged from 0=None to 5=Severe, were higher scores indicated worse pain.
Time Frame: 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 240 | 120
Participants | 174 | 53

5. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Flare.
Description: A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens will be performed without pupil dilation. Scattering of a slit lamp light beam when directed into the anterior chamber (Tyndall effect). The grades for flare were 0=None to 4=Very Severe effect. Complete resolution was defined as Grade 0.
Time Frame: 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 240 | 120
Participants | 152 | 46

6. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells and Flare.
Description: Anterior chamber (AC) cells were assessed using a 0 to 4 grading scale by an ophthalmologist using slip lamp biomicroscopy. A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens was performed without pupil dilation. Accumulation of white blood cells in aqueous was assessed. The grades were defined as: 0 = No cells seen; 1 = 1 - 5 cells; 2 = 6 - 15 cells; 3 = 16 - 30 cells; 4 = >30 cells. Complete resolution of AC cells was defined as Grade 0.
  Anterior Chamber Flare: A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens will be performed without pupil dilation. Scattering of a slit lamp light beam when directed into the anterior chamber (Tyndall effect). The grades for flare were 0=None to 4=Very Severe effect. Complete resolution was defined as Grade 0.
Time Frame: 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 240 | 120
Participants | 67 | 21

7. Secondary Outcome: Percentage of Treatment Failures
Description: Treatment failure was defined as anterior chamber (AC) cell score worsened or remained the same, and the Investigator deemed it necessary to place the participant on rescue therapy.
  Anterior chamber (AC) cells were assessed using a 0 to 4 grading scale by an ophthalmologist using slip lamp biomicroscopy. A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens was performed without pupil dilation. Accumulation of white blood cells in aqueous was assessed. The grades were defined as: 0 = No cells seen; 1 = 1 - 5 cells; 2 = 6 - 15 cells; 3 = 16 - 30 cells; 4 = >30 cells. Complete resolution of AC cells was defined as Grade 0.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 240 | 120
Participants | 17 | 23

ADVERSE EVENTS:
Time Frame: 18 days
Arm/Group | Mapracorat | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/240 | 0/120
Other Adverse Events (participants affected / at risk) | 8/240 | 7/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mapracorat (N=240) | Vehicle (N=120)
Macular edema (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mapracorat (N=240) | Vehicle (N=120)
Eye pain (Eye disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.